CLINICAL TRIAL: NCT06694298
Title: A Phase I Clinical Study of BCMA Chimeric Antigen Receptor T Cell（SYS6020）Injection in Refractory Active Systemic Lupus Erythematosus Patients
Brief Title: A Study of SYS6020 Injection in Refractory Active Systemic Lupus Erythematosus
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYS6020-003
Record Dates: First submitted 2024-11-14; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Refractory Active Systemic Lupus Erythematosus

STUDY DESIGN:
Intervention Model Description: Single Group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SYS6020 (Experimental)
  Interventions: Drug: SYS6020

INTERVENTIONS:
Drug: SYS6020 — BCMA Chimeric Antigen Receptor T Cell（SYS6020）Injection Intravenous infusion
  Other Names: BCMA Chimeric Antigen Receptor T Cell（SYS6020）Injection

SUMMARY:
This study aimed to observe the safety and tolerability of SYS6020 in adult participants with refractory active systemic lupus erythematosus, determine the recommended dose (RD) that may be explored for subsequent studies, and preliminly evaluate the clinical efficacy of this product,and explore the pharmacokinetics and immunogenicity of SYS6020 injection in those participants.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥18 years old, ≤70 years old;
* 2. SLE is diagnosed according to SLICC 2012 or EULAR/ACR 2019 revised criteria.
* 3. Patients are required to have received glucocorticoid combined with immunosuppressive agents and/or biological agents for more than 3 months, with a stable dose for more than 2 weeks, and the disease is still in an active state.
* 4. Antinuclear antibody, anti-ds-DNA antibody and/or anti-Smith antibody are positive.
* 5. SLEDAI-2K score≥7.
* 6. BILAG2004 meets one of the following two criteria:a）BILAG grade A is defined as ≥1 organ system；b）BILAG grade B is defined as ≥2 organ systems
* 7. PGA > 1.0;

Exclusion Criteria:

* 1. Severe lupus nephritis within 8 weeks before screening;
* 2. SLE or non-SLE-related central nervous system disease or lesion within 8 weeks before screening;
* 3. uncontrolled lupus crisis within 8 weeks before screening;
* 4. clinically significant central nervous system diseases or pathological changes other than lupus before screening;
* 5. vasculitis or inflammatory arthritis or skin disease other than SLE or at screening;
* 6. complicated with other autoimmune diseases;
* 7. A B-cell-targeting agent have been used or is planned to be used within 8 weeks before screening，
* 8. received Renal Replacement Therapy（RRT）within 3 months before the screening period or anticipates the need for RRT during the study period;
* 9. participants who will undergo major surgery or invasive intervention within 4 weeks prior to apheresis or plan for systemic or local tumor resection during the study period;
* 10. participants with a known allergy, hypersensitivity, intolerance, or contraindications to SYS6020 or any component of the drugs that may be used in the study,
* 11. active bacterial, fungal, or viral infection within 2 weeks before apheresis;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-12-26 (Estimated); Primary Completion 2029-01-29 (Estimated); Study Completion 2029-01-29 (Estimated)

PRIMARY OUTCOMES:
The frequency and nature of DLT and the incidence of all adverse events and serious adverse events | 28 days after infusion
  Assess safety and tolerability of SYS6020 in patients with systemic lupus erythematosus
recommended dose (RD) | 6 Months
  recommended dose (RD)
Proportion of participants who achieved systemic lupus erythematosus remission (DORIS). | 6 Months
  Proportion of participants who achieved systemic lupus erythematosus remission (DORIS) at 6 months.

SECONDARY OUTCOMES:
Proportion of participants who achieved systemic lupus erythematosus remission (DORIS) | 12 weeks
  Proportion of participants who achieved systemic lupus erythematosus remission (DORIS)
Proportion of participants with complete reduction of hormone dose | 6 Months
  Proportion of participants with complete reduction of hormone dose
Proportion of participants taking ≤5mg/ day of hormone | 6 Months
  Proportion of participants taking ≤5mg/ day of hormone
Proportion of participants achieving low disease activity status (LLDAS) | 12weeks、6 Months
  Proportion of participants achieving low disease activity status (LLDAS)
Absolute and percentage changes from baseline in SLEDA1-2K, BILAG-2004 and PGA scores | 6 Months
  Absolute and percentage changes from baseline in SLEDA1-2K, BILAG-2004 and PGA scores
Changes from baseline in antinuclear antibody, anti-ds-DNA antibody, anti-Smith antibody, C3, C4, and 24-hour urinary protein | 6 Months
  Changes from baseline in antinuclear antibody, anti-ds-DNA antibody, anti-Smith
Changes of immunoglobulin (IgG, IgM, IgA, IgE) from baseline | 6 Months
  Changes of immunoglobulin (IgG, IgM, IgA, IgE) from baseline
Change from baseline in SF-36 | 6 Months
  Change from baseline in SF-36
BCMA CAR+ gene copy numberCAR gene copies | 6 Months
  BCMA CAR+ gene copy numberCAR gene copies
Number of CAR+ cells | 6 Months
  Number of CAR+ cells
Incidence of all adverse events and serious adverse events | 6 Months
  Incidence of all adverse events and serious adverse events